CLINICAL TRIAL: NCT01953211
Title: LH, FHS, Estradiol and Progesterone Activity During the 7-Day Hormone-Free Interval of Various Combined Oral Contraceptive Regimens
Brief Title: Oral Contraceptive Hormone-free Interval Pituitary/ Ovarian Activity
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Frank Stanczyk, Professor, University of Southern California
Other Study IDs: Hormone free interval
Record Dates: First submitted 2013-09-17; First posted 2013-09-30 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Hypothalamic-pituitary-ovarian Axis, Gonadotropins, Ethinyl Estradiol, Contraceptive Efficacy
MeSH Terms: interventions — Contraceptives, Oral, Combined; Ethinyl Estradiol-Norgestrel Combination; norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination; Norinyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy reproductive age women: These volunteers were previously taking the oral contraceptives of interest for a minimum of 3 months
  Interventions: Drug: combined oral contraceptives

INTERVENTIONS:
Drug: combined oral contraceptives
  Other Names: ALESSE, LOESTRIN, NORDETTE, ORTHOCEPT, ORTHOCYCLEN, ORTHO NOVUM

SUMMARY:
The degree of suppression and subsequent activation of the hypothalamic-pituitary-ovarian axis during the hormone-free interval in combined oral contraceptive (COC) hormone users varies depending on the dose of ethinyl estradiol in the formulation. This variation in activation may be associated with different side effects during the hormone free interval. Progesterone (P) remained suppressed during all 6 COC regimens (<1.8 ng/mL), which indicates continuous contraceptive efficacy during the 7-day hormone free interval of all formulations studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, reproductive age women
* 18 to 35 years old,
* seeking contraception from the general gynecology clinics of the LAC and USC Medical Center w
* taking one of 6 possible monophasic COC formulations for at least 3 cycles prior to enrollment
* regular menstrual cycles prior to COCs

Exclusion Criteria:

* Irregular bleeding
* bilateral oophorectomy
* amenorrhea
* hormone-sensitive cancer
* concurrent medications known to interfere with steroid metabolism (i.e., barbiturates, phenytoin, carbamazepine, ethosuximide, primidone, rifampin, tetracycline)

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Healthy, reproductive age women 18 to 35 years old, who were seeking contraception from the general gynecology clinics of the LAC and USC Medical Center were recruited. The research team identified potential candidates who were taking one of 6 possible monophasic COC formulations. Informed consent was obtained from participants by the research staff. To be eligible for participation, women reported regular menstrual cycles prior to COCs, and had taken at least 3 cycles of the same monophasic COC prior to enrollment.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Primary Completion 1998-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LAC and USC Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: clinic
Pre-assignment Details: voluntary
Groups:
- Healthy Reproductive Age Women: These volunteers were previously taking the oral contraceptives of interest for a minimum of 3 months
  combined oral contraceptives
Period: Overall Study
Arm/Group | Healthy Reproductive Age Women
Started | 64 (completed prior to clinical trials submission)
Completed | 64 (completed prior to clinical trials submission)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Reproductive Age Women
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Follicle-stimulating Hormone
Description: mean FSH on day 7 of the pill free interval
Time Frame: Serum blood samples were collected for hormone measurements at the same time daily during the 7 day hormone free interval.
Population: Of note 1 person from the 20 and another from the 30 mcg EE groups hand significant loss of sample and poor processing due to limitations with processing and transport. As a result of this not all participants were able to contribute data for analysis
Measure: Mean (Standard Deviation); unit: milli international units per milliliter
Groups:
- 20 mcg EE; 30 mcg EE; 35 mcg EE: These volunteers were previously taking the oral contraceptives of interest for a minimum of 3 months
Arm/Group | 20 mcg EE | 30 mcg EE | 35 mcg EE
Number analyzed (Participants) | 21 | 21 | 20
milli international units per milliliter | 5.01 (0.25) | 5.86 (0.55) | 6.38 (0.60)
Statistical Analysis 1: Comparison: 20 mcg EE; Test type: Superiority or Other; p = 0.88, t-test, 2 sided; Slope = 0.02, Standard Deviation 0.57
Statistical Analysis 2: Comparison: 30 mcg EE; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Slope = 0.63, Standard Deviation 0.9
Statistical Analysis 3: Comparison: 35 mcg EE; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Slope = 0.83, Standard Deviation 0.78

ADVERSE EVENTS:
Arm/Group | Healthy Reproductive Age Women
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No